CLINICAL TRIAL: NCT00106717
Title: Effectiveness of Narrative Medicine on Pain Intensity and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javeriana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1736
Record Dates: First submitted 2005-03-29; First posted 2005-03-30 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2005-03

CONDITIONS: Cancer
Keywords: Cancer pain; Quality of life; Narrative medicine; Pain relief
MeSH Terms: conditions — Neoplasms; Cancer Pain; Narrative Medicine

INTERVENTIONS:
Procedure: Narrative medicine

SUMMARY:
Narrative medicine addresses the therapeutic benefits that derive from patients forming and telling their personal stories. It offers an innovative model for improving health outcomes. When a patient with cancer and marked suffering writes a narrative of what he or she is going through, this process may reduce pain and improve quality of life.

Therefore, we seek to evaluate the effectiveness of writing a narrative on pain intensity and health related quality of life.

We propose a randomized single blind (evaluator) controlled trial. Patients with cancer pain of intensity at least 5/10 with a minimum Karnofsky score of 50% will be randomized into three groups: 1. Narrative group. Patients will write a story about their illness for at least 20 minutes once a week for 3 weeks; 2. Writing-control group. Patients will fill a pain diary once a week for three weeks; 3. Control group. Subjects will not write/fill anything. Pain will be evaluated using the numerical scale before randomization and then weekly for 8 weeks. We will also evaluate how pain interferes with general activity, mood, work, relation with others, sleep, and enjoyment of life using the Brief Pain Inventory. As secondary outcomes, we will evaluate health related quality of life, with the treatment outcomes of pain survey, which is a modification of the SF 36 (short form health survey), and a global measure of well-being before randomization, and then at 4 and 8 weeks. We will also evaluate the emotional disclosure of the narratives.

We will use an intention to treat analysis. To analyze the effect of the treatment on pain intensity, quality of life, and well-being, we will employ an analysis of repeated measures using generalized estimating equations. We will include in the regression models the treatment group, the emotional disclosure score, the time, and the interaction between treatment group and time.

DETAILED DESCRIPTION:
Background and Significance: To our knowledge there are no randomized controlled trials (RCTs) that evaluate the benefits of narrative medicine, but there has been research on the effect of writing about traumatic events on health outcomes which resembles writing a narrative. However, the populations included have been almost exclusively young healthy students or workers, and the majority of studies have been performed by the same research group.

Study Population: We will recruit patients with cancer who report a pain intensity of at least 5/10. We will include patients who are still able to read and write. To evaluate this physical ability, we will use the Karnofsky scale. The minimum score a patient needs to have will be 50%.

Study Design: This is a randomized single blind (evaluator) controlled trial. Patients will sign an informed consent. Patients will be randomized into three groups.

1. Narrative group. Patients will write a story about their illness for at least 20 minutes once a week for 3 weeks; 2. Writing-control group. Patients will fill a pain diary (requiring approximately 20 minutes) once a week for three weeks; 3. Control group. Subjects will not write/fill out anything.

Patients in the narrative group will be asked to write about their illness and how it has affected their lives. We will not guide the narrative in any other way.

The number of office visits will be the same in the three groups; all patients will be seen weekly up to a total of 8 weeks. In addition, the pain physician will fill a check list to make sure that the presence and severity of symptoms important to patients, such as pain, nausea, anorexia, constipation, and lack of sleep are addressed in all subjects.

We will evaluate the content of the narratives. For the evaluation of the narratives, we will use a Likert scale that goes from no emotional disclosure to very much emotional disclosure. We will also count the number of cognitive words and the number of positive and negative emotion words. The quantitative analysis of vocabulary will be performed with a text-analysis computer program.

Primary Outcome: Reduction of pain intensity is the primary outcome. Pain intensity will be evaluated by a registered nurse, who is not aware of the group allocation, before randomization and then weekly for 8 weeks. To evaluate pain, we will use the numerical rating scale in which 0 is no pain and 10 is the worst pain imaginable.

Secondary Outcomes: Health related quality of life and the sense of well-being are secondary outcomes. For the evaluation of health related quality of life, we will employ the treatment outcomes of pain survey (TOPS) which is a modification of the SF-36 for patients with pain. Patients will fill the questionnaire with the help of a registered nurse, who is not aware of the group allocation, before randomization, and then at 4 weeks and 8 weeks.

For the evaluation of global well-being, we will use a Likert scale that goes from very bad to excellent. Patients will be asked the global measure of well-being weekly.

In addition, we will evaluate how pain interferes with general activity, mood, work, relation with others, sleep, and enjoyment of life using the interference factors of the Brief Pain Inventory (BPI).

Adherence to Treatment: We will call all participants once a week to remind them about writing the story, the pain dairy, or to come to the office visits.

Data Analysis: We will use an intention to treat analysis.

To analyze the effect of the treatment on pain intensity, we will employ an analysis of repeated measures using generalized estimating equations (GEE).

To determine the effect of the exposure on quality of life, we will follow the same procedure described above. The outcome of interest will be the score of each dimension evaluated in the TOPS. As explanatory variables, we will include in the regression models the treatment group, the time, and the interaction between treatment group and time.

To analyze the effect of the exposure on pain interference, we will employ GEE (similar to the procedure we described above). The outcome of interest will be the BPI global score, which is a sum of the scores of each one of the dimensions evaluated (general activity, mood, work, relation with others, sleep, and enjoyment of life). If the BPI global score is different among groups, we then proceed to evaluate each dimension separately to determine which one is affected by narrative medicine. As explanatory variables, we will include in the regression models the treatment group, the time, and the interaction between treatment group and time.

To determine the effect of the exposure on the global measure of well-being, we will use a similar approach described for pain intensity and quality of life. The outcome variable will be the well-being score and the explanatory variables will be treatment group, the time, and the interaction between treatment group and time.

To determine the impact of the quality of the narrative on each of the outcomes evaluated (pain intensity, pain interference, quality of life, and well-being) we will include in the corresponding regression model, in addition to the explanatory variables (treatment group, the time, the interaction between treatment group and time), the emotional disclosure score.

Due to the subjectivity of the emotional disclosure evaluation, two physicians will perform the evaluation (the pain physician and the psychiatrist). We will measure the agreement between the two evaluators using the Kappa statistics for ordinal variables.

To identify and characterize those patients who best respond to narrative medicine, we will include in all the regression models described above the gender, education level, age of the subject, and the interaction between these variables and the treatment group. The evaluation of the interactions will permit us to determine if the effect of narrative medicine depends on the gender, education level, or age of the patients. In addition, we will use latent growth curve analyses to explore the effect of these variables.

To establish the feasibility of narrative intervention, we will compare the number of patients who adhere to the treatment in each group using a chi square test.

Study Period: The exposure will have a duration of 3 weeks and then we will continue the follow up for 5 more weeks, for a total of 8 weeks. We estimate that in 12 months we can finish the recruitment and follow up of the patients and that we need 3 more months to analyze the data and to prepare the manuscript for publication.

Sample Size: We have shown that a difference of 2 units in a scale from 0 to 10 is clinically important to patients. To detect such difference between the groups with 80% power and an alpha error of 0.05, assuming that the baseline pain intensity in our patients will be on average 6 ± 4, we estimated the need for 63 patients per group. To allow for a 10% loss of follow up, we will include a total of 70 patients per group.

To assure that patients with advanced cancer will be similarly distributed in the three groups, we will use a stratified randomization. Our measure of disease severity will be the Karnofsky scale. The cutoff will be 80%. A score of 80% or higher indicates that the patient is able to work.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer pain of intensity at least 5/10 with a minimum Karnofsky score of 50%

Exclusion Criteria:

* Patients unable to write or read

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2004-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity

SECONDARY OUTCOMES:
Pain interference with general activity, mood, work, relation with others, sleep, and enjoyment of life.
Health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: M. Soledad Cepeda, MD, PhD, Principal Investigator — Javeriana University School of Medicine
Locations (1):
- San Ignacio Hospital, Bogotá, DC, Colombia